CLINICAL TRIAL: NCT06800677
Title: Methylated Biomarkers Predictive of Endometrial Cancer Risk
Acronym: BioMEC
Status: Active, not recruiting | Type: Observational
Sponsor: University of Manchester (Other)
Collaborators: Queen Mary University of London (Other)
Responsible Party: Principal Investigator, Sarah Kitson, Clinical Lecturer, University of Manchester
Other Study IDs: 334940
Record Dates: First submitted 2024-07-31; First posted 2025-01-30 (Actual); Last update posted 2025-01-30 (Actual); Status verified 2024-07

CONDITIONS: Endometrial Cancer
Keywords: risk; prevention; prediction
MeSH Terms: conditions — Endometrial Neoplasms | interventions — Hysterectomy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood, urine, cervicovaginal swab, endometrial biopsy, FFPE blocks from hysterectomy specimen including endometrial tumour and normal endometrium
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Cases: Women diagnosed with endometrial cancer of any grade, stage and histological type
  Interventions: Procedure: Hysterectomy
- Controls: Women undergoing a hysterectomy for benign indications
  Interventions: Procedure: Hysterectomy

INTERVENTIONS:
Procedure: Hysterectomy — Elective hysterectomy

SUMMARY:
The goal of this observational study is to identify endometrial cancer risk predictive biomarkers and to optimise the methodology for their detection and quantification in non-invasive samples.

ELIGIBILITY:
Inclusion Criteria:

1. Women aged 45-70 years
2. Attending St Mary's Hospital, Manchester for an elective hysterectomy by any route for either the treatment of endometrial cancer or a benign gynaecological condition
3. Able to consent to participation in the study

Exclusion Criteria:

1. Presence of malignancy asides from endometrial cancer
2. Undergoing elective hysterectomy for suspected ovarian cancer

Ages: 45 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Presence of uterus
Study Population: Women undergoing an elective hysterectomy at St Mary's Hospital, Manchester, UK for either endometrial cancer or a benign indication
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2024-07-31 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Sensitivity, specificity, negative and positive predictive value of single gene methylation classifiers in predicting the presence of endometrial cancer in minimally- and invasive samples | 1 day

SECONDARY OUTCOMES:
Sensitivity, specificity, positive and negative predictive value of a multi-gene methylation classifier for predicting the presence of endometrial cancer | 1 day

CONTACTS AND LOCATIONS:
Locations (1):
- Manchester University NHS Foundation Trust, Manchester, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided
Researchers to write to CI requesting IPD. Fully anonymised data may be shared with other researchers upon receipt of approval from relevant ethics committee